CLINICAL TRIAL: NCT04386876
Title: Randomized, Single Oral Dose,Two Treatment,Four-period,Full-replicated,Cross-over Trial to Assess the BE of Orvical 200 mg/50 mg FT in Comparison With Kaletra 200 mg/50 mg FT in Healthy Male Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Lopinavir/Ritonavir 200/50 mg Film Tablet (World Medicine Ilac, Turkey) Under Fasting Conditions
Acronym: Orvical
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: World Medicine ILAC SAN. ve TIC. A.S. (Industry)
Collaborators: Novagenix Bioanalytical Drug R&D Center (Network); Farmagen Ar-Ge Biyot. Ltd. Sti (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NOV2020/01911; FARGE365 (Other: Farmagen)
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-11

CONDITIONS: Bioequivalence
Keywords: COVID-19 drug treatment; Ritonavir; Lopinavir; Antiviral Agents; Kaletra; Novagenix; Farmagen
MeSH Terms: interventions — Lopinavir; Ritonavir; Motion Pictures; lopinavir-ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Single Oral Dose,Two Treatment,Four-period,Full-replicated,Cross-over
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orvical-Kaletra-Orvical-Kaletra (Experimental): In first and third periods of the study, participants received Orvical 200 mg/50 mg Film Tablet manufactured by World Medicine-Turkey. In second and fourth periods, they received Kaletra 200 mg/50 mg Film CoatedTablet manufactured by AbbVie Deutschland GmbH & Co.-Germany. All periods were performed under fasting state.
  Interventions: Drug: Lopinavir/Ritonavir 200 mg/50 mg Film Tablet; Drug: Lopinavir/Ritonavir 200 mg/50 mg Film Coated Tablet
- Kaletra-Orvical-Kaletra-Orvical (Experimental): In first and third periods of the study, participants received Kaletra 200 mg/50 mg Film Coated Tablet manufactured by AbbVie Deutschland GmbH & Co.-Germany. In second and fourth periods, they received Orvical 200 mg/50 mg Film Tablet manufactured by World Medicine-Turkey. All periods were performed under fasting state.
  Interventions: Drug: Lopinavir/Ritonavir 200 mg/50 mg Film Tablet; Drug: Lopinavir/Ritonavir 200 mg/50 mg Film Coated Tablet

INTERVENTIONS:
Drug: Lopinavir/Ritonavir 200 mg/50 mg Film Tablet — Lopinavir/Ritonavir film tablet containing 200 mg lopinavir and 50 mg ritonavir (World Medicine-Turkey).
  Other Names: Orvical 200 mg/50 mg Film Tablet
Drug: Lopinavir/Ritonavir 200 mg/50 mg Film Coated Tablet — Lopinavir/Ritonavir film coated tablet containing 200 mg lopinavir and 50 mg ritonavir(AbbVie Deutschland GmbH & Co.-Germany)
  Other Names: Kaletra 200 mg/50 mg Film Coated Tablet

SUMMARY:
A single dose of Reference product containing 200 mg lopinavir and 50 mg ritonavir fixed dose combination and a single dose of Test product containing 200 mg lopinavir and 50 mg ritonavir fixed dose combination or vice versa; administered with 240 mL of water at room temperature, in each period under fasting conditions.

DETAILED DESCRIPTION:
The subjects will me isolated at the dorm during 5 days before the dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian male subjects aged between 20 and 40 years,
2. Non smokers or smoking maximum 5 cigarettes a day, those who won't smoke or drink coffee during the study period,
3. Negative Covid-19 Rapid Test results and two Negative Covid-19 PCR test results,
4. Negative alcohol breath test results,
5. Normal physical examination at screening visit,
6. Having the Body Mass Index ranged between 18.5-30 kg/m2 (see Appendix I) which is in the desirable range according to the age,
7. Ability to communicate adequately with the investigator himself or his representatives,
8. Ability and agreement to comply with the study requirements,
9. Normal blood pressure and heart rate measured under stabilised conditions at the screening visit after at least 5 minutes of rest under supine position: SBP within 100 to 140 mmHg, DBP within 60 to 90 mmHg and HR within 50 to 90 bpm,
10. Normal/ acceptable 12-lead electrocardiographic results at least after 5 minutes of rest,
11. Laboratory results within normal range or clinically non-significant (CBC, glucose, urea, uric acid, creatinine, estimated GFR (eGFR), total bilirubin, sodium, potassium, calcium, chloride, SGOT (AST), SGPT (ALT), GGT, alkaline phosphatase, total protein and urinalysis), drug addiction scanning in urine results in negative (amphetamine, barbiturate, benzodiazepine, cannabinoid, cocaine, opiate),
12. Understanding of the study and agreement to give a written informed consent according to section 20.3.
13. Volunteer's compliance with isolation rules defined at study protocol

Exclusion Criteria:

1. Who have atopic constitution or asthma or known allergy for lopinavir and ritonavir or any other ingredients of the products.
2. Any history or presence of clinical relevance of cardiovascular (myocardial infarction/ ischaemia and/or QT prolongation etc.), neurological, musculoskeletal, haematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease, any type of porphyria.
3. Baseline ECG should be performed at screening. Exclude subjects having a QTc > 440 ms
4. Symptomatic or asymptomatic orthostatic hypotension at screening or before the first drug administration defined by a decrease of SBP more than 20 mmHg or DBD more than 10 mmHg occurs between sitting/supine to standing position subject will be excluded (if it deemed necessary by the investigator),
5. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
6. Subjects who have given more than 400 mL blood within the last two months before the first drug administration and subjects who have participated to any drug research within the last two months before the first drug administration.
7. Subjects suspected to have a high probability of non-compliance to the study procedure and/or completion of the study according to the investigator's judgement.
8. Subjects who used any of prescribed systemic or topical medication (including OTC medication) within 2 weeks (or six elimination half lives of this medication, whichever is longer) before the initiation of the study (except single doses of analgesics which have no drug interaction with study product).
9. Use of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
10. Subjects who have any chronic disease which might interfere with absorption, distribution, metabolism or excretion of the drug.
11. Subjects who regular consumed of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine, chocolate, sodas,) equivalent to more than 500 mg methylxanthines per day.
12. Subjects who has taken any grapefruit or grapefruit juice during 7 days prior to drug administration, during the study.
13. History of allergic response to heparin.
14. History of drug abuse.
15. History of alcohol abuse and/or regular use of more than 2 units of alcohol per day or 10 units per week and/or positive alcohol breath test results (Note: one unit of alcohol equals 250 mL beer, 125 mL wine or 25 mL spirits).
16. Positive blood test for HBV, HCV and HIV.
17. Who have relationship to the investigator.
18. Who are not suitable to any of inclusion criteria.
19. History of difficulty of swallowing.
20. Intake of depot injectable solutions (including study medications) within 6 months before start of the study.
21. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before start of the study.
22. Special diet due to any reason, e.g. vegetarian.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Primary PK End Points | 12 weeks
  AUC0-tlast of lopinavir and ritonavir
Primary PK End Points | 13 weeks
  Cmax of lopinavir and ritonavir

CONTACTS AND LOCATIONS:
Overall Officials: Muradiye Nacak, MD,PhD, Principal Investigator — Farmagen Ar-Ge Biyot. Ltd. Sti
Locations (2):
- Turkey (Türkiye) (2):
  - Novagenix Drug R&D Center, Akyurt, Ankara
  - Farmagen Ar-Ge Biyot. Ltd. Sti., Şahinbey, Gaziantep

DOCUMENTS (2):
  • Informed Consent Form (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT04386876/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT04386876/Prot_SAP_001.pdf